CLINICAL TRIAL: NCT03779854
Title: Multi-Center Phase II Randomized Controlled Trial of Naïve T Cell Depletion for Prevention of Chronic Graft-Versus-Host Disease in Children and Young Adults
Brief Title: Naive T Cell Depletion for Preventing Chronic Graft-versus-Host Disease in Children and Young Adults With Blood Cancers Undergoing Donor Stem Cell Transplant
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RG1003345; 9880 (Other: Fred Hutch/University of Washington Cancer Consortium); NCI-2018-01752 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); P30CA015704 (NIH); RG1003345 (Other: Fred Hutch/University of Washington Cancer Consortium); P01CA018029-43 (NIH)
Record Dates: First submitted 2018-12-17; First posted 2018-12-19 (Actual); Last update posted 2025-10-15 (Actual); Status verified 2025-10

CONDITIONS: Acute Biphenotypic Leukemia; Acute Leukemia; Acute Leukemia of Ambiguous Lineage; Acute Lymphoblastic Leukemia; Acute Undifferentiated Leukemia; Allogeneic Hematopoietic Stem Cell Transplantation Recipient; Blastic Plasmacytoid Dendritic Cell Neoplasm; Blasts Under 25 Percent of Bone Marrow Nucleated Cells; Blasts Under 5 Percent of Bone Marrow Nucleated Cells; Mixed Phenotype Acute Leukemia; Myelodysplastic Syndrome With Excess Blasts-1; Myelodysplastic Syndrome/Acute Myeloid Leukemia; Burkitt Leukemia; Chronic Monocytic Leukemia; Lymphoblastic Lymphoma; Mast Cell Leukemia; Myeloproliferative Neoplasm
MeSH Terms: conditions — Leukemia, Biphenotypic, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Blastic Plasmacytoid Dendritic Cell Neoplasm; GATA2 Deficiency; Burkitt Lymphoma; Leukemia, Myeloid; Leukemia, Mast-Cell; Myeloproliferative Disorders | interventions — Whole-Body Irradiation; Thiotepa; fludarabine; fludarabine phosphate; Cyclophosphamide; Busulfan; Bone Marrow Transplantation; Tacrolimus; Methotrexate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm I (chemotherapy, naive T-cell depleted PBSC) (Experimental): CONDITIONING REGIMEN A: Patients undergo TBI BID on days -10 to -7, then receive thiotepa IV over 3 hours QD on days -6 and -5, and fludarabine IV over 30 minutes once daily on days -6 to -2.
  CONDITIONING REGIMEN B: Patients undergo TBI BID on days -8 to -5, then receive fludarabine IV over 30 minutes QD on days -4 to -2, and cyclophosphamide IV over 1 hour QD on days -3 and -2.
  CONDITIONING REGIMEN C: Patients receive fludarabine IV over 30 minutes QD on days -6 to -2, busulfan IV over 180 minutes QD on days -5 to -2, and undergo total body irradiation BID on day -1.
  TRANSPLANT: Patients receive naive T-cell depleted PBSCs on day 0.
  GVHD PROPHYLAXIS: All patients receive tacrolimus IV beginning on day -1 and methotrexate IV on days 1, 3, 6, and 11.
  Additionally, patients undergo ECHO and CSF collection at baseline as well as blood sample collection and bone marrow aspiration with or without biopsy throughout the trial.
  Interventions: Radiation: Total-Body Irradiation; Drug: Thiotepa; Drug: Fludarabine; Drug: Cyclophosphamide; Drug: Busulfan; Drug: Tacrolimus; Drug: Methotrexate; Procedure: Naive T Cell-Depleted Hematopoietic Stem Cell Transplantation; Procedure: Echocardiography; Procedure: Biospecimen Collection; Procedure: Bone Marrow Aspiration; Procedure: Bone Marrow Biopsy
- Arm II (chemotherapy, unmanipulated T cell replete BM) (Active Comparator): CONDITIONING REGIMEN A: Patients undergo TBI BID on days -10 to -7, then receive thiotepa IV over 3 hours QD on days -6 and -5, and fludarabine IV over 30 minutes once daily on days -6 to -2.
  CONDITIONING REGIMEN B: Patients undergo TBI BID on days -8 to -5, then receive fludarabine IV over 30 minutes QD on days -4 to -2, and cyclophosphamide IV over 1 hour QD on days -3 and -2.
  CONDITIONING REGIMEN C: Patients receive fludarabine IV over 30 minutes QD on days -6 to -2, busulfan IV over 180 minutes QD on days -5 to -2, and undergo total body irradiation BID on day -1.
  TRANSPLANT: Patients receive unmanipulated T cell-replete BM on day 0.
  GVHD PROPHYLAXIS: All patients receive tacrolimus IV beginning on day -1 and methotrexate IV on days 1, 3, 6, and 11.
  Additionally, patients undergo ECHO and CSF collection at baseline as well as blood sample collection and bone marrow aspiration with or without biopsy throughout the trial.
  Interventions: Radiation: Total-Body Irradiation; Drug: Thiotepa; Drug: Fludarabine; Drug: Cyclophosphamide; Drug: Busulfan; Procedure: Allogeneic Bone Marrow Transplantation; Drug: Tacrolimus; Drug: Methotrexate; Procedure: Echocardiography; Procedure: Biospecimen Collection; Procedure: Bone Marrow Aspiration; Procedure: Bone Marrow Biopsy

INTERVENTIONS:
Radiation: Total-Body Irradiation — Undergo TBI
  Other Names: Total Body Irradiation; Whole-Body Irradiation; SCT_TBI; TBI; Whole Body Irradiation
Drug: Thiotepa — Given IV
  Other Names: 1,1',1"-phosphinothioylidynetrisaziridine; Oncotiotepa; STEPA; Tepadina; Tespamin; Tespamine; Thio-Tepa; Thiofosfamide; Thiofozil; Thiophosphamide; Thiophosphoramide; triethylenethiophosphoramide
Drug: Fludarabine — Given IV
  Other Names: 2-Fluoro-9-beta-arabinofuranosyladenine; 2-Fluorovidarabine; Fluradosa
Drug: Cyclophosphamide — Given IV
  Other Names: Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; Cycloblastin; Cytophosphane
Drug: Busulfan — Given IV
  Other Names: Bussulfam; Busulfanum; Busulfex; Busulphan; Misulban; Misulfan; Mitosan; Myeleukon
Procedure: Allogeneic Bone Marrow Transplantation — Receive unmanipulated T cell replete BM
  Other Names: Allo BMT; Allogeneic Blood and Marrow Transplantation; Allogeneic BMT
  Arms: Arm II (chemotherapy, unmanipulated T cell replete BM)
Drug: Tacrolimus — Given IV
  Other Names: Fujimycin; Hecoria; Prograf; Protopic
Drug: Methotrexate — Given IV
  Other Names: Abitrexate; Alpha-Methopterin; Amethopterin; Brimexate; Emtexate; Emthexat; Emthexate; Farmitrexat; Medsatrexate; Methoblastin; Rheumatrex
Procedure: Naive T Cell-Depleted Hematopoietic Stem Cell Transplantation — Receive naive T-cell depleted PBSCs
  Arms: Arm I (chemotherapy, naive T-cell depleted PBSC)
Procedure: Echocardiography — Undergo ECHO
  Other Names: EC; ECHO
Procedure: Biospecimen Collection — Undergo CSF and blood sample collection
Procedure: Bone Marrow Aspiration — Undergo bone marrow aspiration
Procedure: Bone Marrow Biopsy — Undergo bone marrow biopsy

SUMMARY:
This phase II trial studies how well naive T-cell depletion works in preventing chronic graft-versus-host disease in children and young adults with blood cancers undergoing donor stem cell transplant. Sometimes the transplanted white blood cells from a donor attack the body's normal tissues (called graft versus host disease). Removing a particular type of T cell (naive T cells) from the donor cells before the transplant may stop this from happening.

DETAILED DESCRIPTION:
Patients are randomized to 1 of 2 arms. All patients receive 1 of 3 conditioning regimens.

CONDITIONING REGIMEN A: Patients undergo total body irradiation (TBI) twice daily (BID) on days -10 to -7, then receive thiotepa intravenously (IV) over 3 hours once daily (QD) on days -6 and -5, and fludarabine IV over 30 minutes once daily on days -6 to -2.

CONDITIONING REGIMEN B: Patients undergo TBI BID on days -8 to -5, then receive fludarabine IV over 30 minutes QD on days -4 to -2, and cyclophosphamide IV over 1 hour QD on days -3 and -2.

CONDITIONING REGIMEN C: Patients receive fludarabine IV over 30 minutes QD on days -6 to -2, busulfan IV over 180 minutes QD on days -5 to -2, and undergo total body irradiation BID on day -1.

ARM I: Patients receive naive T-cell depleted PBSCs on day 0.

ARM II: Patients receive unmanipulated T cell-replete BM on day 0.

GVHD PROPHYLAXIS: All patients receive tacrolimus IV on days -1 to +50 followed by a taper in the absence of grade II-IV aGVHD. Patients also receive methotrexate IV on days +1, +3, +6, and +11.

Additionally, all patients undergo echocardiography (ECHO) and cerebrospinal fluid (CSF) collection at baseline as well as blood sample collection and bone marrow aspiration with or without biopsy throughout the trial.

After completion of study treatment, patients are followed up at days 28, 56, 90, 180, 270, and 365 and then at months 15, 18, 21, and 24.

ELIGIBILITY:
Inclusion Criteria:

* The patient must have one of the following diagnoses and be considered to be an appropriate candidate for allogeneic HCT by the study site principal investigator (PI):

  * Acute lymphoblastic leukemia (ALL) with < 5% marrow blasts.
  * Acute myeloid leukemia (AML) with < 25% marrow blasts.
  * Other acute leukemia (OAL) or related neoplasm (including but not limited to acute biphenotypic leukemia [ABL], ambiguous lineage [ALAL], mixed phenotype acute leukemia [MPAL], blastic plasmacytoid dendritic cell neoplasm [BPDCN], acute undifferentiated leukemia [AUL], lymphoblastic lymphoma, Burkitt leukemia/lymphoma, mast cell leukemia, chronic monocytic leukemia [CML] with blast crisis or other chronic myeloproliferative neoplasm) with < 5% marrow blasts.
  * Myelodysplastic syndrome (MDS) with excess blasts (EB-1 and EB-2) and has received cytotoxic induction chemotherapy (excluding small molecule inhibitors and de-methylating agents)
* Age 6 months to 26 years at the time informed consent is obtained using the Informed Consent to Participate in a Research Study form
* Matched related donor (MRD) or matched unrelated donor (MUD) (defined as 8/8 match for human leukocyte antigen [HLA]-A, -B, -C, -DRB1).
* Planned product type for infusion is PBSC or BM (i.e. not cord blood):

  * For feasibility phase, planned product type for infusion must be PBSC.
  * For RCT, planned product type must be PBSC or BM.
* Karnofsky or Lansky score >= 60%.
* Left ventricular ejection fraction (LVEF) at rest >= 40%.
* Diffusing capacity of the lungs for carbon monoxide (DLCO) (corrected for hemoglobin) >= 60% predicted by pulmonary function tests (PFTs)

  * Patients who are unable to perform PFTs (age < 6 years or considered developmentally incapable of PFTs): oxygen saturation (by oximetry) must be >= 92% on room air.
* Total bilirubin =< 2 x upper limit of normal (ULN) (unless value[s] > 2 x ULN are disease- or medication-related).

  * If value(s) are > 2 x ULN and not disease- or medication related, patient must be evaluated by a gastrointestinal (GI) physician. If GI physician considers protocol treatment to be contraindicated for the patient, the patient will not be eligible for the study.
* Alanine aminotransferase (ALT), aspartate aminotransferase (AST) =< 2 x ULN (unless value[s] > 2 x ULN are disease- or medication-related).

  * If value(s) are > 2 x ULN and not disease- or medication related, patient must be evaluated by a gastrointestinal GI physician. If GI physician considers protocol treatment to be contraindicated for the patient, the patient will not be eligible for the study.
* Serum creatinine (SCr) within normal range for age. If SCr is outside normal range for age, creatinine clearance (CrCl) > 40 mL/min/1.73m^2 must be obtained (measured by 24-hour [hr] urine specimen or nuclear glomerular filtration rate [GFR]).

  * Age (Years): Maximum SCr (mg/dL)
  * =< 5: 0.8
  * 6-10: 1
  * 11-15: 1.2
  * > 15: 1.5
* Recipient informed consent/assent/legal guardian permission documentation must be obtained.
* DONOR: May be related (MRD) or unrelated (MUD) to the subject.
* DONOR: Must be matched to the subject at 8/8 HLA alleles (HLA-A, -B, -C, and -DRB1)
* DONOR: Be >=14 years of age.
* DONOR: Must be available to donate in the United States of America (USA) (i.e. excludes international donors).
* DONOR: Must agree to donate BM or PBSC (i.e. agree to donate whichever product type is requested) (applicable only to the RCT phase of this study).
* DONOR: MUDs:

  * Must give informed consent according to applicable National Marrow Donor Program (NMDP) donor regulatory requirements
  * Must meet eligibility criteria as defined by the NMDP or be ineligible with statement of urgent medical need (exception 21 CFR 1271.65(b)(iii))

    * Tests must be performed using Food and Drug Administration (FDA) licensed, cleared, and approved test kits in a Clinical Laboratory Improvement Amendments (CLIA)-certified laboratory
* DONOR: MRDs:

  * Must be negative for human immunodeficiency virus (HIV)-1, HIV-2, human T-lymphotropic virus (HTLV)-1, HTLV-2, hepatitis B, hepatitis C (serological and/or nucleic acid testing [NAT] and/or other approved testing)
  * Must meet institutional donor eligibility criteria, or be ineligible with statement that the donor is a first or second degree relative (exception 21 CRF 1271.65(b)(i)).

    * Tests must be performed using FDA licensed, cleared, and approved test kits in a CLIA-certified laboratory.

Exclusion Criteria:

* Active central nervous system (CNS) disease. A patient may have a history of CNS disease; however, any CNS disease must be cleared by the end of the pre-conditioning evaluation. If CNS disease is identified on the first cerebrospinal fluid (CSF) evaluation within 30 days of the start of the preparative regimen, a repeat CSF evaluation must be performed and show no evidence of disease in order for the patient to be eligible for the protocol.
* Patients on other experimental protocols for the prevention of GVHD.
* Patient body weight:

  * Matched related donor (MRD): > 100 kg are ineligible
  * Matched unrelated donor (MUD): > 75 kg must be discussed with the protocol principal investigator (PI) prior to enrollment.
* HIV-positive.
* Uncontrolled infections must be evaluated by an infectious disease physician and considered suitable to undergo HCT by the study site PI, infectious disease physician and protocol PI. Upper respiratory tract infection (URI) does not constitute an uncontrolled infection in this context.
* Life expectancy < 3 months from disease other than acute leukemia or myelodysplastic syndrome (MDS).
* Significant medical condition that would make recipient unsuitable for HCT.
* Prior allogeneic or autologous HCT.
* Females who are pregnant or breastfeeding.
* Patients of child bearing age who are presumed to be fertile and are unwilling to use an effective birth control method or refrain from sexual intercourse during study treatment and for 12 months following HCT.
* Known hypersensitivity to tacrolimus, fludarabine, or methotrexate (MTX).

Ages: 6 Months to 26 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 68 (Estimated)
Dates: Start 2019-08-29 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Feasibility achievement | Up to 2 years
  Success defined as achievement of cell selection goals for two consecutive Naive T cells (TN)-depleted peripheral blood stem cells (PBSC) hematopoietic cell transplantation (HCTs) at each study site (Feasibility)
Engraftment of neutrophils by day 28 (Feasibility) | At day 28
  Success defined as achievement neutrophil engraftment (absolute neutrophil count [ANC] >= 500/mm^3) on first day of three consecutive laboratory values obtained on different days.
Current-graft versus host disease (GVHD)-free, relapse-free survival (Randomized Controlled Trial [RCT]) | At 1 year
  Defined as alive, no relapse after HCT, no current GVHD requiring prednisone, no graft rejection or graft failure. The proportion of subjects meeting the primary endpoint will be described in each arm with 90% confidence intervals (CI) and compared between arms using the chi-square test. A two-sided 10% significance level will be used for this comparison.

SECONDARY OUTCOMES:
Chronic GVHD (cGVHD) meeting National Institutes of Health (NIH) criteria and requiring prednisone (RCT) | At 1 and 2 years
  Cumulative incidence curve will be computed for each arm along with a 90% CI at 1 year and 2 years post-HCT. Death and/or relapse prior to occurrence of cGVHD will be considered as competing risks. The cumulative incidence curves will be compared between arms using Gray's test. The maximum severity of cGVHD will also be described in each arm and compared using the chi-squared test.
Proportion of subjects alive and off prednisone (or equivalent systemic corticosteroid) for treatment of GVHD (RCT) | At 3, 6, 9, 12, 15, 18, 21 and 24 months post HCT
  Proportions of subjects alive without requiring use of prednisone (or equivalent systemic corticosteroid) for GVHD will be estimated with 90% CI for both arms at time points over 24 months, and compared using the chi-squared test.

CONTACTS AND LOCATIONS:
Overall Officials: Marie Bleakley, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (10):
- United States (10):
  - Children's Hospital of Los Angeles, Los Angeles, California
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Children's Healthcare of Atlanta, Atlanta, Georgia
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - Dana Farber / Boston Children's Hospital, Boston, Massachusetts
  - UH Rainbow Babies and Children's Hospital (University Hospitals Cleveland Medical Center), Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bleakley M. Naive T-cell depletion in stem cell transplantation. Blood Adv. 2020 Oct 13;4(19):4980. doi: 10.1182/bloodadvances.2020001888. PMID 33049057